CLINICAL TRIAL: NCT02074371
Title: Perioperative Parameters to Predict Postoperative Respiratory Depression After Cardiac Surgery
Brief Title: Postoperative Respiratory Depression After Cardiac Surgery
Acronym: CABG PRD
Status: Completed | Type: Observational
Sponsor: Ovidiu Constantin Baltatu (Other)
Responsible Party: Sponsor-Investigator, Ovidiu Constantin Baltatu, Professor, Universidade Camilo Castelo Branco
Organization: Universidade Camilo Castelo Branco (Other)
Other Study IDs: BR-002-SJC; CEP-UESP128/11 (Other: UESP)
Record Dates: First submitted 2014-02-26; First posted 2014-02-28 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery bypass surgery; cardiopulmonary bypass; ICU; postoperative respiratory depression
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Coronary artery bypass graft surgery (CABG) is associated with postoperative respiratory depression. In this study we aimed at investigating perioperative parameters that could predict the nadir of postoperative respiratory function impairment.

DETAILED DESCRIPTION:
Coronary artery bypass graft (CABG) surgery is a principal revascularization option for ischemic heart disease and the principal modality for invasive treatment of coronary artery disease. Postoperative pulmonary complications are the most frequent and significant contributor to length of hospitalization, morbidity and mortality. The objective of this study is to search for perioperative parameters that could predict the degree of impairment of respiratory function after CABG with cardiopulmonary bypass (CPB).

ELIGIBILITY:
Inclusion Criteria:

* patients of both sexes older than 18 years submitted to CABG with CPB, presence of coronary disease confirmed by coronary angiography, use of the left internal thoracic artery and/or saphena, patients who remained in spontaneous ventilation on the first postoperative day, absence of chronic or acute pulmonary disease, and giving written informed consent to participate in the study.

Exclusion Criteria:

* intraoperative change of the surgical technique, surgical complications or complications occurring in the ICU, emergency reoperation, renal failure, failure to agree to continue in the study, presence of other types of heart disease, and presence of pulmonary diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease submitted to elective CABG with CPB.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Postoperative Respiratory Depression After Cardiac Surgery | 9 days
  Respiratory function is assessed through maximal inspiratory (MIP) and expiratory (MEP) pressures and peak expiratory flow (PEF) determined 1 day before surgery and one postoperative week.

SECONDARY OUTCOMES:
Intraoperative parameters after coronary artery bypass graft surgery (CABG) | 1 day
  Intraoperative parameters are monitored, including volume of cardioplegia, CPB duration, aortic cross-clamp time, number of grafts.
Perioperative parameters after coronary artery bypass graft surgery (CABG) | 3 days
  ICU blood pressure is monitored

CONTACTS AND LOCATIONS:
Overall Officials: Ovidiu C Baltatu, MD PhD, Study Chair — Camilo Castelo Branco University (UNICASTELO)
Locations (1):
- Hospital Sao Marcos, Teresina, Piauí, Brazil

REFERENCES:
- [Derived] Costa AS, Costa PH, de Lima CE, Padua LE, Campos LA, Baltatu OC. ICU Blood Pressure Variability May Predict Nadir of Respiratory Depression After Coronary Artery Bypass Surgery. Front Neurosci. 2016 Jan 11;9:506. doi: 10.3389/fnins.2015.00506. eCollection 2015. PMID 26903799
- See also: Published data — http://journal.frontiersin.org/article/10.3389/fnins.2015.00506/full?utm_source=Email_to_authors_&utm_medium=Email&utm_content=T1_11.5e1_author&utm_campaign=Email_publication&field=&journalName=Frontiers_in_Neuroscience&id=165510